CLINICAL TRIAL: NCT01092793
Title: Effect of Superba Krill on Inflammation in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Krill-2010
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2010-03

CONDITIONS: Stable Atherosclerotic Coronary Disease
Keywords: Fish oil; Krill; CAD
MeSH Terms: interventions — krill protein extract; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Krill (Active Comparator)
  Interventions: Dietary Supplement: Krill
- Fish oil (Active Comparator)
  Interventions: Dietary Supplement: Fish oil
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Krill — Encapsulated oil from the antarctic crustacean Krill
  Arms: Krill
Dietary Supplement: Fish oil — Encapsulated, raffined cod-oil
  Arms: Fish oil

SUMMARY:
Atherosclerotic coronary heart disease is a condition thought to involve low-grade inflammation. Several reports, clinical and epidemiological, have demonstrated that intake of fish oil may be beneficial in attenuating the inflammatory process. Still, however, there are lacking data in respect to whether differences in composition of various marine oils may influence the inflammatory status differently.

The hypothesis of the current study is that extract from the antarctic krill (Euphausia superba) is better than traditional fish oils when compared head-to-head with balanced composition of omega 3 content on inflammatory status.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years
* Sex: Male and female
* Stable atherosclerotic coronary heart disease (heart attack >3 months ago or objectified angina pectoris).
* No hospitalization for heart disease last 3 months.

Exclusion Criteria:

* Unstable heart disease.
* Heart failure NYHA class III and IV.
* Previous valve and/or aortic surgery
* Significant concomitant disease (i.e. diseases with known inflammatory activation - e.g. various autoimmune diseases, chronic infections, significant acute infections three weeks before or during the study, connective tissue disease, arthritis, chronic pulmonary disease or serious liver- or kidney-disease).
* Simultaneous involvement in other clinical studies involving intervention.
* Planned operation or other invasive procedures (e.g. PCI etc.) during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Inflammatory blood status | 8 weeks intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Oslo University Hospital / Rikshospitalet, Oslo, Norway